CLINICAL TRIAL: NCT03441191
Title: Audio-visual Stimulation for Sleep Promotion in Older Adults With Osteoarthritis Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Jean Tang, Assistant Professor, Nursing: Department Of Psychosocial And Community Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 48538
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Insomnia Chronic; Osteoarthritis; Pain, Chronic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Osteoarthritis; Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active AVS (Experimental): Active AVS consists of a 30-minute pulsing lights (red, green, blue) and sounds that gradually descend from alpha (10 Hz) to delta (2 Hz).
  Interventions: Device: Audiovisual Stimulation
- Placebo Control AVS (Placebo Comparator): The placebo control AVS program consists of 30 minutes of constant dim light that slowly changes in color, and a steady monotone at ultra-low (<1 Hz) frequency (outside of the entrainment range).
  Interventions: Device: Audiovisual Stimulation

INTERVENTIONS:
Device: Audiovisual Stimulation — A commercially available AVS device (MindPlace Procyon) modified for use in the current study will be used to deliver the AVS programs in this study

SUMMARY:
Background and Purpose: The purpose of the study is to test the efficacy of an audio-visual stimulation program for sleep promotion in adults with chronic pain. The hypothesis is that hyper-arousal plays an important role in insomnia. Brainwave entrainment from 8 to 1 Hz reduces arousal, and thereby improves sleep. Improved sleep may change how people perceive pain.

Methods: Using a double-blind, randomized controlled trial design, we plan to enroll 30 adults (21-65 years old) experiencing both nonmalignant pain and insomnia. Exclusion criteria include: seizure disorder, sleep disorder, and night shift workers. After a one-week baseline measure, participants will be randomized to intervention or placebo group. Participants in both groups will be asked to self-administer the audio-visual stimulation program every night at bedtime for one month. Upon completion, post intervention measures will be collected.

DETAILED DESCRIPTION:
Background: The purpose of this pilot study was to test the efficacy of an open-looped Audio-visual Stimulation program (AVS) for sleep promotion in older adults with osteoarthritis pain. In this study, the AVS program was tested in a randomized controlled design. Specifically, this pilot study examined a 30-minute audio-visual stimulation program that gradually ramped from 10 Hz down to 2 Hz, to be used at bedtime for delta brainwave induction, in a randomized controlled design. The placebo control AVS program consisted of 30-minutes of constant dim light that slowly changed in color, and a steady monotone at ultra-low (<1 Hz) frequency (outside of the entrainment range).

Method: A total of 30 older adults (mean age 68 ± 5.1, 90% women) with comorbid insomnia and osteoarthritis pain participated in this 2-week study. Participants were randomly assigned to either AVS active program or AVS placebo control program. After the baseline assessment (which included questionnaires [sleep, pain, depression], and quantitative electroencephalogram (QEEG) during AVS induction), participants were asked to self-administer their group specific AVS program nightly at bedtime for two weeks. Post-treatment questionnaires (sleep, pain, depression) were then collected.

ELIGIBILITY:
Inclusion Criteria:

* 60 years or older
* Having difficulty sleeping over the past three months (Insomnia Severity Index ≥ 8)
* Having osteoarthritis pain (Brief Pain Inventory Worst pain ≥ 4)

Exclusion Criteria:

* Working night shift
* Previously diagnosed with a primary sleep disorder (Sleep Apnea or Restless Leg Syndrome).
* Seizure disorder
* Photosensitivity
* Dementia
* Diagnosis or other significant chronic illness beyond OA that would impact sleep
* Severe psychiatric disorder including a history of or current diagnosis of psychosis

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2016-11-01 (Actual)

PRIMARY OUTCOMES:
Insomnia of Severity Index | 2 weeks post baseline
  A 7-item questionnaire that is a global measure of perceived insomnia severity. Items use a 5-point scale for total scores of 0-28, with >15 considered moderate severity. The ISI has good internal consistency and is sensitive to changes in sleep of older adults in clinical and research.
Pittsburgh Sleep Quality Index (PSQI) | 2 weeks post baseline
  Self-rating of overall sleep quality and disturbances using 7 sleep components. A PSQI global score >5 is highly sensitive and specific for distinguishing good and poor sleepers.
Brief Pain Inventory (BPI) short form | 2 weeks post baseline
  The BPI is a 9-item questionnaire that assesses severity of pain, impact of pain on daily function, location of pain, pain medications and amount of pain relief in the past 24 hours or the past week.

SECONDARY OUTCOMES:
Patient Health Questionnaire | 2 weeks post baseline
  The PHQ-9 is a 9-item reliable, valid, measure that rates depression symptom severity on a 4-point scale.
Sleep Diary | baseline through 2 weeks post baseline
  The sleep diary is a two-page sleep log with standard fill in the blank questions about the quantity and quality of the previous night of sleep, including Time to Bed, Sleep Latency, Number of Awakenings, Wake After Sleep Onset time, Total Sleep Time, and Time out of Bed. The diary also includes questions about the causes of sleep difficulties and ratings of daytime fatigue and sleepiness.
Actigraphy | baseline through 2 weeks post baseline
  Sleep and wake pattern (actigraph) will be measured by Philips Respironics Actiwatch-2. Actigraphy is a reliable and objective tool to monitor sleep-wake cycles in ambulatory individuals (including older adults) based on frequency and magnitude of movements.
Quantitative Electroencephalogram (QEEG) | baseline
  Cortical activity will be evaluated using a 19-channel quantitative electroencephalographic system (Discovery 24E, BrainMaster)30 with a standard electrode cap that has 22 sensors attaching to the scalp.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Tang, PhD, Principal Investigator — University of Washington

REFERENCES:
- [Background] Tang HY, Vitiello MV, Perlis M, Riegel B. Open-Loop Neurofeedback Audiovisual Stimulation: A Pilot Study of Its Potential for Sleep Induction in Older Adults. Appl Psychophysiol Biofeedback. 2015 Sep;40(3):183-8. doi: 10.1007/s10484-015-9285-x. PMID 25931250
- [Background] Tang HY, Vitiello MV, Perlis M, Mao JJ, Riegel B. A pilot study of audio-visual stimulation as a self-care treatment for insomnia in adults with insomnia and chronic pain. Appl Psychophysiol Biofeedback. 2014 Dec;39(3-4):219-25. doi: 10.1007/s10484-014-9263-8. PMID 25257144
- [Background] Tang HY, Riegel B, McCurry SM, Vitiello MV. Open-Loop Audio-Visual Stimulation (AVS): A Useful Tool for Management of Insomnia? Appl Psychophysiol Biofeedback. 2016 Mar;41(1):39-46. doi: 10.1007/s10484-015-9308-7. PMID 26294268